CLINICAL TRIAL: NCT03782805
Title: Effect of Vitamin D Treatment on Some Inflammatory Markers in Non-obese Lebanese Patients With Type 2 Diabetes
Brief Title: Effect of Vitamin D Supplementation on Inflammatory Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 222222
Record Dates: First submitted 2018-12-13; First posted 2018-12-20 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Vitamin D Deficiency; Type2 Diabetes
Keywords: vitamin D, type 2 diabetes, inflammation
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes Mellitus, Type 2; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: In this randomized, controlled, double blind study, participants were randomized (using the simple randomization method) to receive either a supplement of 10,000 IU of cholecalciferol (Euro-Pharm International, Canada) or a placebo tablet (containing microcrystalline cellulose: 66.3%, starch: 33.2%, magnesium stearate: 0.5%, per serving) to be taken 3 times a week for a period of six months
Who Masked: Participant, Investigator
Masking Description: Neither the investigator nor the subjects were aware of the group allocation; the pharmacist (in charge of the placebo tablets as well as the packing and coding of the supplements) was the only person to know to which group each participant belonged.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Group receiving a supplement of 10,000 IU of cholecalciferol (Euro-Pharm International, Canada) to be taken 3 times a week for a period of six months.
  Interventions: Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)
- Placebo group (Placebo Comparator): Group receiving a placebo tablet (containing microcrystalline cellulose: 66.3%, starch: 33.2%, magnesium stearate: 0.5%, per serving) to be taken 3 times a week for a period of six months
  Interventions: Dietary Supplement: Placebo tablet

INTERVENTIONS:
Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada) — The participants are randomly asked to take either a pill containing either a supplement of cholecalciferol or placebo for 3 times a week, within a period of 6 months
  Arms: treatment group
Dietary Supplement: Placebo tablet — The participants are randomly asked to take either a pill containing either a supplement of cholecalciferol or placebo for 3 times a week, within a period of 6 months
  Arms: Placebo group

SUMMARY:
Previous studies have shown that improving vitamin D status among the elderly may lead to an improvement in some inflammatory markers, especially with patients with type 2 diabetes. The aim of our trial is study the effect of vitamin D supplementation on inflammatory markers in patients having type 2 diabetes.

DETAILED DESCRIPTION:
Vitamin D was shown crucial for insulin secretion and glucose homeostasis. Furthermore, one of the markers of type 2 diabetes is low-grade inflammation, which can be the result of an elevated circulation of cytokines. High amounts of circulating inflammatory cytokines such as tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6) contribute significantly to insulin resistance in muscle and adipose tissues. The aim of this randomized, controlled, double blind study is to examine the effect of vitamin D supplementation on some inflammatory markers in older Lebanese patients having type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects deficient in vitamin D
* Subjects having type 2 diabetes
* Non-obese subjects

Exclusion Criteria:

* Subjects having hyperparathyroidism
* Subjects suffering from hepatic disease / kidney disease

Ages: 60 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline fasting blood glucose (FBG) at 6 months | baseline and after 6 months of intervention
  FASTING BLOOD GLUCOSE
Change from Baseline Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at 6 months | baseline and after 6 months of intervention
  Homeostatic Model Assessment of Insulin Resistance
Change from Baseline C-reactive protein (CRP) at 6 months | baseline and after 6 months of intervention
  C-reactive protein
Change from Baseline Interleukin-6 (IL-6) at 6 months | baseline and after 6 months of intervention
  Interleukin-6
Change from Baseline TNF-alpha at 6 months | baseline and after 6 months of intervention
  TNF-alpha

SECONDARY OUTCOMES:
Change from Baseline weight at 6 months | baseline and after 6 months of intervention
  weight change
Change from Baseline Body Mass Index (BMI) at 6 months | baseline and after 6 months of intervention
  Body mass index
Change from Baseline waist circumference at 6 months | baseline and after 6 months of intervention
  Waist circumference change
Change from Baseline Percentage of fat at 6 months | baseline and after 6 months of intervention
  Percentage of fat
Change from Baseline Parathyroid hormone (PTH) at 6 months | baseline and after 6 months of intervention
  Parathyroid hormone

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia E Hajj, PhD, Study Director — Dr
Locations (1):
- Saint Charles Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
The plan will be shared upon request

REFERENCES:
- [Background] Yu Y, Tian L, Xiao Y, Huang G, Zhang M. Effect of Vitamin D Supplementation on Some Inflammatory Biomarkers in Type 2 Diabetes Mellitus Subjects: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Ann Nutr Metab. 2018;73(1):62-73. doi: 10.1159/000490358. Epub 2018 Jun 26. PMID 29945132
- [Background] Safarpour P, Vafa MR, Amiri F, Janani L, Noorbakhsh M, Rajabpour Nikoo E, Sadeghi H. A double blind randomized clinical trial to investigate the effect of vitamin D supplementation on metabolic and hepato-renal markers in type 2 diabetes and obesity. Med J Islam Repub Iran. 2018 Apr 28;32:34. doi: 10.14196/mjiri.32.34. eCollection 2018. PMID 30159285
- [Derived] El Hajj C, Walrand S, Helou M, Yammine K. Effect of Vitamin D Supplementation on Inflammatory Markers in Non-Obese Lebanese Patients with Type 2 Diabetes: A Randomized Controlled Trial. Nutrients. 2020 Jul 9;12(7):2033. doi: 10.3390/nu12072033. PMID 32659891